CLINICAL TRIAL: NCT02271542
Title: Identification of Polymorphisms Involved in the Metabolism of Propofol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayse Ulgey, Resident, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2013/215
Record Dates: First submitted 2014-10-19; First posted 2014-10-22 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: UGT1A1*28 Polymorphism
Keywords: Propofol; Polymorphism; UGT1A9; CYP2B6
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- between 1-10 ages (Experimental): Propofol, 1-2 mg / kg after the installation is 100 to 200 mg / kg / min infusion for 30-60 minutes after application will be made and EDTA tubes with 2 ml blood sample will be taken. Determined from blood samples obtained by studying the polymorphism genotypes of patients will be exposed.
  Interventions: Drug: propofol
- under 60 ages (Experimental): Propofol, 1-2 mg / kg after the installation is 100 to 200 mg / kg / min infusion for 30-60 minutes after application will be made and EDTA tubes with 2 ml blood sample will be taken. Determined from blood samples obtained by studying the polymorphism genotypes of patients will be exposed.
  Interventions: Drug: propofol
- upper 60 ages (Experimental): Propofol, 1-2 mg / kg after the installation is 100 to 200 mg / kg / min infusion for 30-60 minutes after application will be made and EDTA tubes with 2 ml blood sample will be taken. Determined from blood samples obtained by studying the polymorphism genotypes of patients will be exposed.
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: propofol — Propofol, 1-2 mg / kg after the installation is 100 to 200 mg / kg / min infusion for 30-60 minutes after application will be made and EDTA tubes with 2 ml blood sample will be taken. Determined from blood samples obtained by studying the polymorphism genotypes of patients will be exposed.
  Other Names: pofol

SUMMARY:
Identification of Polymorphisms Involved in the Metabolism of Propofol

DETAILED DESCRIPTION:
Propofol inside and outside the operating room during anesthesia is a drug widely used. In terms of efficacy and side effect profile of propofol knows if properties are insufficient data on the metabolism. Propofol typically undergoes biotransformation by microsomal enzymes in the liver. For most of the administered dose, takes place glucuronidation by UGT1A9 enzyme, while the remaining portion is oxidized with CYP2B6 hydroxylation reactions. However, these enzymes are involved in the metabolism of propofol are enzymes highly polymorphic. Polymorphisms occurring in these enzymes; the effects of propofol, side effects and drug needs to show individual differences in terms of causes. Determination of the genetic background of individuals and personal anesthetic regimen improved. Thus, useful person drug resistance, increased incidence of side effects can be reduced. In particular, be aware of some mutations, such as propofol infusion syndrome mortal side effects can be prevented. The main purpose of this study, these individual differences are thought to be the cause of polymorphic variation in UGT1A9 and CYP2B6 gene to determine. Especially in the UGT1A9 gene mutations that may be associated with ethnic structure can be observed. In Caucasian, African-American communities and polymorphisms of this gene has been shown in Japanese. So all of them as a result of the genetic structure of any society can be considered as its own. Therefore, this study aimed to determine the genetic polymorphism of Turkish society has.Physiological factors such as age and sex between persons of different answers to the causes of propofol. Another object of this study was the identification of these factors can lead to different answers which is to present the relationship between polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who used propofol for induction onl
* Between the ages of 1-85

Exclusion Criteria:

* Patients taking drugs that may affect the metabolism of propofol (exp.Ketamine)
* Smoking and Alcohol users
* Patients using herbal medicines

Ages: 1 Year to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Polymorphism | 60 minutes after induction
  EDTA blood samples from patients for the study of polymorphisms, DNA will be obtained with the help of DNA isolation kit. DNA isolation from blood samples taken after the sample is stored at -80 ° C until the operating phase.
  Research priorities included in the appropriate primers for each polymorphism will be created.
  Using appropriate PCR program, will be determined the genotype of each polymorphism.

CONTACTS AND LOCATIONS:
Overall Officials: Halil AKBULUT, Resident, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No